CLINICAL TRIAL: NCT01184482
Title: A Phase I Study of Lapatinib and Cetuximab in Patients With Solid Tumors
Brief Title: Lapatinib and Cetuximab in Patients With Solid Tumors
Acronym: TYKERB-ITUX 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tykerb-itux 1; 2010-218 (Other: Georgetown University)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Colorectal Cancer; Lung Cancer; Head and Neck Cancer
Keywords: recurrent colorectal cancer; recurrent head and neck cancer; recurrent lung cancer; cetuximab; lapatinib
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Head and Neck Neoplasms | interventions — Cetuximab; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab and lapatinib (Experimental): All patients will receive cetuximab by IB weekly and daily doses of lapatinib orally in 3 week cycles with response assessed every 2 cycles.
  Interventions: Drug: cetuximab and lapatinib

INTERVENTIONS:
Drug: cetuximab and lapatinib — Cetuximab: 400 mg/m2 on Day 1 then 250 mg/m2 weekly
  Lapatinib: Start once daily on Day 1. Dose escalating cohorts:
  1. 750 mg (3 tabs)
  2. 1000 mg (4 tabs)
  3. 1250 mg (5 tabs)
  Other Names: Cetuximab: erbitux; Lapatinib: tykerb

SUMMARY:
This trial is for patients with colon cancer, head and neck cancer and lung cancer that has not responded to standard therapy.

Cetuximab targets a receptor on cancer cells called the Epidermal Growth Factor Receptor or EGFR. It is thought that this receptor is turned "on" in some cancers, enabling cancer cells to divide and grow. Blocking this receptor can turn this signal off. Cetuximab blocks this receptor from the outside of cancer cells. It is thought that cancer cells can turn this signal back on by the EGFR joining with a related receptor called ErbB2. Lapatinib blocks both EGFR and ErbB2 from the inside of cancer cells. In laboratory experiments it has been found that combining drugs that target both EGFR and ErbB2 might work better in turning this signal back off. The purpose of this study is to determine the maximum dosages that patients can tolerate when these two medicines are given at the same time.

In addition, in order to be on this trial, patients must agree to have a tumor biopsy before starting treatment on this study and 21 days after starting treatment. These biopsies are a required part of the study. Patients must also agree to have blood drawn for research testing to see whether genetic differences between patients explain different reactions to and side effects from, these medicines.

ELIGIBILITY:
Inclusion Criteria:

* At least one measurable lesion by RECIST criteria
* A tumor lesion that can be readily biopsied using a core needle via clinical exam, ultrasound, CT, or fluoroscopic-guidance
* Over the age of 18 years and able to provide informed consent
* Patients must have progressed after standard therapy for metastatic/ recurrent disease including 5-FU containing regimens for patients with colorectal cancer, and platinum-containing regimens for patients with head and neck cancer and non-small cell lung cancer.
* Patients may have received cetuximab, panitumumab or erlotinib previously
* Adequate kidney, liver, and bone marrow function
* Life expectancy greater than 3 months
* ECOG performance status </= 2
* Normal left ventricular ejection fractions

Exclusion Criteria:

* Chemotherapy or surgery within 4 weeks prior to treatment start
* Radiation treatment within 3 weeks prior to treatment start
* Prior therapy with lapatinib
* Untreated brain metastasis or neurologically unstable CNS metastases
* Any severe or uncontrolled medical condition or other condition that could affect participation in this study including unstable angina, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction </= 6 months prior to study entry
* Diarrhea > grade 1 at baseline
* Patients on a medication or herbal therapy known to inhibit CYP3A4
* Gastrointestinal tract disease resulting in the inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption or active peptic ulcer disease
* Ongoing ventricular cardiac dysrhythmias of grade >/= 2
* Subjects with a history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation >= 3 beats in a row)
* Serious cardiac arrhythmia requiring medication
* QTc interval > 500 msec
* Female patients who are pregnant or breast feeding, or adults who are of reproductive potential and are unwilling to refrain from conceiving a child during study treatment
* Patients unwilling or unable to comply with the protocol or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 12 months
  The dose at which </= 1 out of 6 subjects experiences a dose limting toxicity

SECONDARY OUTCOMES:
response rate | 12 months
  How well tumor responds to treatment as measured by RECIST criteria
Pharmacokinetics | 12 months
  Pharmacokinetics of lapatinib as measured by weekly trough levels
Genetic polymorphisms | 12 months
  genetic polymorphisms in ABCG2, ABCB1, CYP3A4, and CYP3A5 wil be identified and counted
Genetic variations and activation status for EGFR and ErbB2 pathways | 12 months
  Genetic variations and activation status for EGFR amd ErbB2 pathways will be measured in pre- and post-therapy biopsies and assessed with western blots and IHC.

CONTACTS AND LOCATIONS:
Overall Officials: John F Deeken, M.D., Principal Investigator — Georgetown Univeristy Medical Center
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States